CLINICAL TRIAL: NCT01970969
Title: This Study Will Investigate the Association Between a Set of Single Nucleotide Polymorphisms (SNPs) and Atrial Fibrillation in Patients at High Risk of Developing Atrial Fibrillation. The SNPs Investigated Will Have Been Previously Shown to be Associated With the Atrial Fibrillation.
Brief Title: THE GIRAFFE Study: Genomic Risk Markers for Atrial Fibrillation Following Extended Cardiac Rhythm Monitoring
Acronym: GIRAFFE
Status: Completed | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Collaborators: Quest Diagnostics-Nichols Insitute (Industry)
Responsible Party: Sponsor
Other Study IDs: 13-6159
Record Dates: First submitted 2013-10-08; First posted 2013-10-28 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Patients With Symptoms of Cardiac Arrhythmia at Risk for Atrial Fibrillation
Keywords: Atrial Fibrillation; Cardiac monitoring; Genomics
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — A blood sample (in a 4 ml EDTA tube) for genotyping and a serum sample (in two 10ml red top tubes) will be obtained from each patient.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cardiac arrhythmia symptoms: All subjects enrolled in the study will have an iRhythm Zio patch placed and a blood sample obtained.

SUMMARY:
Our primary hypothesis is that a risk score comprised of approximately 10 single nucleotide polymorphisms (SNPs) that are associated with atrial fibrillation at the Genome Wide Association Study (GWAS) level is associated with the development of atrial fibrillation among previously undiagnosed patients at high risk for atrial fibrillation. A current example of these SNPs is shown in Table 1. As a secondary hypothesis, we will test the association between atrial fibrillation diagnosed in this study with a subset of SNPs reported to be associated with atrial fibrillation and with fine-mapping SNPs. We will also test the association between atrial fibrillation of less than and greater than 30 seconds and a panel of approximately 10 SNPs.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of high clinical suspicion for atrial fibrillation prompting referral for ambulatory cardiac rhythm monitoring for potential atrial fibrillation.

AND

* At high risk for atrial fibrillation, defined as any one of the following: ischemic stroke with no defined etiology (In prior 6 months) [3, 4, 6, 7], hypertension [33], increased body mass index (BMI >30kg/m2) [33], heart failure [33], clinically significant murmur [33], prolonged PR interval on resting ECG [33], chronic kidney disease [34], hypertrophic cardiomyopathy [35], congenital heart disease [36], chronic obstructive pulmonary disease [37, 38], sleep apnea [39-41], thyroid disease [42, 43], family history of atrial fibrillation [44], diabetes [45] or excess alcohol consumption (Male > 14 drinks/week, Female >7 drinks/week)[46].
* Age 40 years or older
* Capable of providing informed consent
* Capable of wearing a Zio Patch for up to 14 days
* Capable of providing a blood sample

Exclusion Criteria:

* Previously documented atrial fibrillation or atrial flutter.
* Prior cardiac surgery (coronary artery bypass grafting, valve replacement or repair, pericardial stripping, etc) within the past 30 days.
* Hyperthyroidism.
* Have known skin allergies, conditions, or sensitivities (e.g. allergy to adhesives, psoriasis) as the Zio Patch should not be used on patients with known skin allergies, conditions, or sensitivities.
* Are receiving pacing therapy.
* Are anticipated to receive or require external cardiac defibrillation during the monitoring period.
* Are anticipated to have exposure to high frequency surgical equipment during the monitoring period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients defined, as high risk for atrial fibrillation will be persons with:
  1. No prior history of atrial fibrillation and/or atrial flutter (AFIB/AF) - with symptoms of high clinical suspicion for AFIB/AF prompting referral for ambulatory cardiac rhythm monitoring to evaluate for potential AFIB/AF, and
  2. Any of the following features: ischemic stroke with no defined etiology (In prior 6 months) [3, 4, 6, 7], hypertension [33], increased body mass index (BMI >30kg/m2) [33], heart failure [33], clinically significant murmur [33], prolonged PR interval on resting ECG (>200msec) [33], chronic kidney disease [34], hypertrophic cardiomyopathy [35], congenital heart disease [36], chronic obstructive pulmonary disease [37, 38], sleep apnea [39-41], thyroid disease [42, 43], family history of atrial fibrillation [44], diabetes [45] or excess alcohol consumption (Male > 14 drinks/week, Female >7 drinks/week)[46].
Sampling Method: Non-Probability Sample
Enrollment: 928 (Actual)
Dates: Start 2013-09; Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Association between events of Atrial Fibrillation and 4-SNP risk score | One time
  SNP effect sizes and frequencies were determined from the literature and the International HapMap Project database as indicated in Table 1. Expected occurrences of atrial fibrillation in the two groups were calculated using reference to previous studies as outlined above [7, 8, 33]. We expect 80 atrial fibrillation events in a 650 high-risk patients [48, 49]. Using these event rates and an alpha error of 5%, the power to detect an association between a 10-SNPs risk score and atrial fibrillation is >90%. The power to detect association between a 4-SNP risk score and atrial fibrillation is >80%.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Topol, MD, Principal Investigator — Scripps Translational Science Institute
Locations (1):
- Scripps Clinic, La Jolla, California, United States

REFERENCES:
- [Derived] Muse ED, Wineinger NE, Spencer EG, Peters M, Henderson R, Zhang Y, Barrett PM, Rivera SP, Wohlgemuth JG, Devlin JJ, Shiffman D, Topol EJ. Validation of a genetic risk score for atrial fibrillation: A prospective multicenter cohort study. PLoS Med. 2018 Mar 13;15(3):e1002525. doi: 10.1371/journal.pmed.1002525. eCollection 2018 Mar. PMID 29534064